CLINICAL TRIAL: NCT05465863
Title: Humoral and Cellular İmmune Response to SARS-CoV-2 mRNA BNT162b2 Vaccine in Pediatric Kidney Transplant Recipients Compared to Dialysis Patients and Healthy Children
Brief Title: Humoral and Cellular İmmune Response to SARS-CoV-2 mRNA BNT162b2 Vaccine in Children With Chronic Kidney Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayca Kiykim, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COVIDCKD
Record Dates: First submitted 2022-07-19; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Chronic Kidney Disease 5D; Chronic Kidney Disease 5T
Keywords: children; chronic kidney disease; covid19; vaccination; antibody response
MeSH Terms: conditions — Renal Insufficiency, Chronic; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Active Comparator)
  Interventions: Biological: SARS-CoV-2 mRNA BNT162b2 vaccine (Pfizer-BioNTech®)
- Healthy controls (Active Comparator)
  Interventions: Biological: SARS-CoV-2 mRNA BNT162b2 vaccine (Pfizer-BioNTech®)

INTERVENTIONS:
Biological: SARS-CoV-2 mRNA BNT162b2 vaccine (Pfizer-BioNTech®) — When permitted by local guidelines, children and adolescents who were over 12 years old were notified of vaccine eligibility and encouraged to schedule an appointment

SUMMARY:
Coronavirus 2019 (COVID-19) infection is associated with higher morbidity and mortality in adult patients on dialysis, and kidney transplant recipients (KTRs). Although children had lower morbidity and mortality, KTRs are more vulnerable than healthy children.

It has already known that the general immune responses to vaccines, which are currently in practice (attenuated, conjugated, or recombinant) were lower than healthy controls in children and adolescents on dialysis and with a kidney transplantation. Uremic milieu and immunosuppressive drugs are the factors causing impaired immune response in this group of patients. The new mRNA vaccine technology is used worldwide including children and adolescents during the pandemic. Studies have demonstrated lower immune response to new SARS-CoV-2 mRNA vaccine in adult KTRs. However, there is limited data about vaccine-induced immune response in children and adolescent with renal replacement therapy.

The aim of this study was to assess immune response to SARS-CoV-2 mRNA BNT162b2 and its clinical and laboratory correlates in children and adolescent KTRs. Humoral immune response was assessed by anti-SARS-CoV-2 immunoglobulin G (Anti-S IgG) and its clinical correlate neutralizing antibody (nAb). Cellular immune response was assessed with SARS-CoV-2 specific Interferon ɣ release assay (IGRA).

DETAILED DESCRIPTION:
This is a prospective, multicenter case-control study performed between September 2021 and March 2022 in the Pediatric Nephrology Units of IU- Cerrahpaşa School of Medicine, Memorial Hospital, Marmara University School of Medicine, IU- Istanbul School of Medicine, Medeniyet University School of Medicine, and Istinye University School of Medicine. The control group has consisted of age and gender comparable 19 healthy children without any acute infection or chronic disease, who were admitted to Cerrahpasa School of Medicine, Pediatric out-patient unit for routine control.

When permitted by local guidelines, children and adolescents who were over 12 years old were notified of vaccine eligibility and encouraged to schedule an appointment. The SARS-CoV-2 mRNA BNT162b2 vaccine (Pfizer-BioNTech®) administered to all participants by intramuscular route in the deltoid region. At least one month after the second dose of the vaccine, serum samples and whole blood samples were collected from all patients and controls, to analyze the humoral and cellular immune response to the vaccine. All samples were stored at -20 ◦C until testing. SARS-CoV-2 PCR test results were recorded retrospectively to determine natural infection.

ELIGIBILITY:
Inclusion Criteria:

* 12-21 year-old chronic kidney diseases and dialysis patients

Exclusion Criteria:

* Patients with primary immune deficiencies and not vaccinated with SARS-CoV-2 mRNA BNT162b2 vaccine
* Patients who did not completed 2 series of SARS-CoV-2 mRNA BNT162b2 vaccine

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the antibody response following vaccination | one month after the second dose of the vaccine
  Anti-SARS-CoV-2 IgG Quantification and Neutralisation test

SECONDARY OUTCOMES:
Evaluation of the cellular response following vaccination | one month after the second dose of the vaccine
  Interferon Gamma Release Assay

CONTACTS AND LOCATIONS:
Locations (6):
- Turkey (Türkiye) (6):
  - Istanbul University-Cerrahpasa, Istanbul
  - Istanbul University, Istanbul School of Medicine, Istanbul
  - Istinye University, School of Medicine, Istanbul
  - Marmara University, School of Medicine, Istanbul
  - Medeniyet University, School of Medicine, Istanbul
  - Memorial Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gulmez R, Ozbey D, Agbas A, Aksu B, Yildiz N, Uckardes D, Saygili S, Yilmaz EK, Yildirim ZY, Tasdemir M, Kiykim A, Cokugras H, Canpolat N, Nayir A, Kocazeybek B, Caliskan S. Humoral and cellular immune response to SARS-CoV-2 mRNA BNT162b2 vaccine in pediatric kidney transplant recipients compared with dialysis patients and healthy children. Pediatr Nephrol. 2023 Jul;38(7):2199-2208. doi: 10.1007/s00467-022-05813-w. Epub 2022 Dec 2. PMID 36459243